CLINICAL TRIAL: NCT07264829
Title: COMPARATIVE ANALYSIS OF INTRA-PULPAL CRYOTHERAPY METHODS DURING PULPECTOMY IN MOLARS WITH SYMPTOMATIC IRREVERSIBLE PULPITIS: A RANDOMIZED CONTROL TRIAL
Brief Title: This Randomized Controlled Trial Evaluates the Effectiveness of Two Intra-pulpal Cryotherapy Methods, Endo-ice and Ice Sticks, in Reducing Intra-operative Pain and Improving Anesthesia Success During Pulpectomy of Mandibular Molars With Symptomatic Irreversible Pulpitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tina Lohana, FCPS Resident, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-3725/DUHS/Approval/2024/74
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Root Canal Treatment; Intra-operative Pain; Symptomatic Irreversible Pulpitis; Cryotherapy Effect
Keywords: Cryotherapy; Endodontic treatment; Intra-operative pain; Pulpectomy; Endo-ice; Ice-sticks; Symptomatic Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The principal investigator will perform the endodontic procedure, with the outcome assessor blinded to the cryotherapy method. Prior to administering IANB, a topical anesthetic gel will be applied. A 27-gauge needle will deliver 1.8 ml of 2% lidocaine with 1:100,000 epinephrine at a rate of 1 ml/min. After a 5-minute wait, anesthesia effectiveness will be confirmed through electric pulp testing (EPT) on a neighboring tooth, with two consecutive negative responses confirming success. Once adequate anesthesia is confirmed, an access opening will be made under rubber dam isolation for the procedure.
  In Control Group, after access opening and complete de-roofing of the pulp chamber, pulpectomy of the inflamed pulp will be performed under the given effective Inferior alveolar nerve block with no additional intervention to control intra-operative pain.
- Endo-ice Group (Experimental): The principal investigator will perform the endodontic procedure, with the outcome assessor blinded to the cryotherapy method. Prior to administering IANB, a topical anesthetic gel will be applied. A 27-gauge needle will deliver 1.8 ml of 2% lidocaine with 1:100,000 epinephrine at a rate of 1 ml/min. After a 5-minute wait, anesthesia effectiveness will be confirmed through electric pulp testing (EPT) on a neighboring tooth, with two consecutive negative responses confirming success. Once adequate anesthesia is confirmed, an access opening will be made under rubber dam isolation for the procedure.
  In Endo-ice Group, after access opening, pulp will be exposed and de-roofing will be performed. Endo-ice with the help of cotton pellet will be applied inside the pulp chamber for 2min (8 consecutive applications, 15sec each) and pulpectomy of the inflammed pulp will be performed immediately.
  Interventions: Other: Endo-ice (Refrigerant Spray)
- Ice-sticks Group (Experimental): The principal investigator will perform the endodontic procedure, with the outcome assessor blinded to the cryotherapy method. Prior to administering IANB, a topical anesthetic gel will be applied. A 27-gauge needle will deliver 1.8 ml of 2% lidocaine with 1:100,000 epinephrine at a rate of 1 ml/min. After a 5-minute wait, anesthesia effectiveness will be confirmed through electric pulp testing (EPT) on a neighboring tooth, with two consecutive negative responses confirming success. Once adequate anesthesia is confirmed, an access opening will be made under rubber dam isolation for the procedure.
  In Ice-sticks Group, following the access opening and complete de-roofing of pulp chamber, four ice sticks will be placed inside the pulp chamber for 2 minutes (30 seconds each, using tweezer). Subsequently, pulpectomy of the inflamed pulp will be performed immediately.
  Interventions: Other: Ice-sticks

INTERVENTIONS:
Other: Endo-ice (Refrigerant Spray) — Endo-ice (1,1, 1,2-Tetrafluoroethane, Refrigerant spray) have been most frequently used in dentistry to assess pulp sensibility. In this study, Endo-ice will be used to perform intra-coronal cryotherapy and its effectiveness in reducing intra-operative pain will be evaluated.
  Arms: Endo-ice Group
Other: Ice-sticks — Ice-sticks have been mostly used in dentistry to assess pulp sensibility. In this study, Ice-sticks will be used to perform intra-coronal cryotherapy and it's effectiveness in reducing intra-operative pain will be evaluated.
  Arms: Ice-sticks Group

SUMMARY:
The goal of this clinical trail is to compare the analgesic effect of endo-ice and ice-sticks in reducing intra-operative pain during pulpectomy in molars with Symptomatic Irreversible Pulpitis. Principal Investigator will perform the procedure and outcome assessor will interview the participants as well as fill the pre-operative questionnaire. The patient will be instructed beforehand on how to score their pre-operative, intra-operative and post-operative intensity of pain according to Visual Analogue Scale.The Anxiety level of patient will also be recorded according to the Corah's Dental Anxiety Scale questionnaire and their level of anxiety before and after the intervention will be recorded by the outcome assessor.

The principal investigator will perform all endodontic procedures, with the outcome assessor blinded to the cryotherapy method. Prior to administering IANB, a topical anesthetic gel will be applied. A 27-gauge needle will deliver 1.8 ml of 2% lidocaine with 1:100,000 epinephrine at a rate of 1 ml/min. After a 5-minute wait, anesthesia effectiveness will be confirmed through electric pulp testing (EPT) on a neighboring tooth, with two consecutive negative responses confirming success. Once adequate anesthesia is confirmed, an access opening will be made under rubber dam isolation for the procedure.

1. CONTROL GROUP: After access opening and complete de-roofing of the pulp chamber, pulpectomy of the inflamed pulp will be performed under the given effective IANB with no additional intervention to control intra-operative pain.
2. ENDO-ICE GROUP: After access opening, pulp will be exposed and de-roofing will be performed. Endo-ice with the help of cotton pellet will be applied inside the pulp chamber for 2min (8 consecutive applications, 15sec each) and pulpectomy of the inflammed pulp will be performed immediately.
3. ICE-STICKS GROUP: Following the access opening and complete de-roofing of pulp chamber, four ice sticks will be placed inside the pulp chamber for 2 minutes (30 seconds each, using tweezer). Subsequently, pulpectomy of the inflamed pulp will be performed immediately.

Patients will be asked to rate their level of pain to the outcome assessor at four specific intervals during the trial, i.e., pre-operative (before local anesthesia), pre-operative (after local anesthesia), during pulpectomy and immediately after pulp extirpation and it will be recorded in a proforma by the blinded outcome assessor.

Pain and Anxiety Scores will be compared to asses either cryotherapy or which method of cryotherapy found to be effective in reducing intra-operative pain.

DETAILED DESCRIPTION:
INTRODUCTION:

Acute pain associated with symptomatic irreversible pulpitis (SIP) can be induced by any stimuli or occur spontaneously and may persist for up to 30 seconds or beyond the removal of the stimulus, signaling the need for endodontic treatment. An essential prerequisite for successful endodontic therapy is effective pulpal anesthesia. The standard method for achieving regional anesthesia in mandibular molar involves an inferior alveolar nerve block (IANB) combined with buccal infiltration. However, an IANB does not always provide successful pulpal anesthesia, particularly in patients with symptomatic irreversible pulpitis (SIP).The occurrence of pain during endodontic treatment of teeth with SIP poses a significant challenge for both the clinician and the patient. In such circumstances, painless pulp extirpation becomes challenging. In endodontics, cryotherapy has been used following periradicular surgeries and as a final irrigant (cold saline) before obturation to reduce postoperative pain and inflammation.

METHODOLOGY:

This research will be conducted using a randomized controlled trial at Dow International Dental College. The target demographics includes 60 individuals with pain mandibular molars, experiencing moderate to severe pain (VAS 4-10), diagnosed with symptomatic irreversible pulpitis, planned for endodontic treatment. Pulpal sensibility will be assessed with cold test and electric pulp tester. Digital peri-apical x-rays will be used to evaluate the extent of caries and periapical status. Group allocation will be done by Computer generated random numbers. Individuals will be divided into 3 groups (20 each). 1. Control Group 2. Cryotherapy with endo-ice 3. Cryotherapy with ice-sticks. Cryotherapy methods (Endo-ice and Ice-sticks) will be used as an intervention to control per-operative pain in Intervention Groups and no additional measures will be taken to control pain in Control group, which is the standard method). After confirming the success of anesthesia, procedure will be started in all 3 groups.

The outcome assessor will interview the participants as well as fill the pre-operative questionnaire. The patient will be instructed beforehand on how to score their pre-operative, intra-operative and post-operative intensity of pain according to VAS. Similarly, for anxiety assessment, the patients will be interviewed according to the DAS-R questionnaire and their level of anxiety before and after the intervention will be recorded by the outcome assesor.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals (Male and Female) aged 18 to 40 years.
2. Healthy individuals with no significant present and past medical findings.
3. Mandibular molars.
4. Symptomatic irreversible pulpitis (moderate to severe pain according to VAS 4-10).
5. Periapical index (PAI) Score: 1-3 on periapical radiograph.
6. DAS-R: 4-14( mild to moderate anxiety)

Exclusion Criteria:

1. Immature teeth with open apices.
2. Calcified pulp chamber and canals.
3. Periodontally compromised teeth.
4. Individuals who had taken steroids, analgesics, or antibiotics within the last 48 hours.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Measuring Intra-operative pain using Visual Analogue Scale | 3 hours
  Patient will be interviewed at different intervals during the procedure and pain scores will recorded with the help of Visual Analogue Scale

SECONDARY OUTCOMES:
Measuring Anxiety during procedure using Corah's Dental Anxiety Scale | 3 hours
  Patient will be interviewed by the outcome assessor before and after the procedure and anxiety will be measured using Corah's Dental Anxiety Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Farah Naz, BDS, FCPS, Study Chair — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No